CLINICAL TRIAL: NCT03034681
Title: Lumbosciatic Syndrome: a Quasi-experimental Study on the Effectiveness of the Vojta Therapy vs. Transcutaneous Electrical Nerve Stimulation
Brief Title: Lumbosciatic Syndrome: Vojta Therapy vs. TENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Collaborators: Research Support Unit at Hospital General Mancha Centro (Unknown)
Responsible Party: Principal Investigator, María Lidia Juarez, Physiotherapist and clinical profesor, Universidad Rey Juan Carlos
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 280920168216
Record Dates: First submitted 2017-01-16; First posted 2017-01-27 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Lumbosciatic Syndrome; Pain; Functional Limitation; Vojta Therapy; Transcutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The patients were recruited as follows: the rehabilitation doctor evaluated and diagnosed the patient and referred them to the Physiotherapy Unit (PTU) with a prescription for "TENS or Vojta" treatment. It was at the PTU of the health centre where the patient was informed of the possibility of taking part in the study. Patients who agree were allocated alternately in order of arrival to the PTU, in such a way that half of the sample was treated using TENS and the other half with Vojta therapy .
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vojta (Other): Vojta therapy consists in activating certain overall and innate locomotion patterns or complexes: reflex creeping and reflex rolling, which provokes the contraction of striated muscle in the entire body in a determined coordination with the central nervous system (CNS). These patterns are triggered from different positions (prone, supine and side lying) and only with certain stimulation. They contain all the locomotion components: automatic postural control, uprighting and phase movements. This therapy allows for the changing from pathological patterns to painless and cheaper patterns. This group received 15 sessions of treatment. Treatment lasted 30 minutes per sesion.
  Interventions: Other: Physiotherapy technique: Vojta Therapy
- TENS (Active Comparator): TENS procedure used at our unit consists in applying a high frequency current (80Hz), which is the most effective way to combat pain, for a phase duration of 60-200 microseconds at a comfortable range. Electrodes are placed on the skin over the sciatic nerve path, the (-) cathode on the most painful area as it is the most stimulating and the (+) another is placed distal. This group received 15 sessions of treatment. Treatment lasted 30 minutes per sesion.
  Interventions: Other: Physiotherapy technique: TENS

INTERVENTIONS:
Other: Physiotherapy technique: TENS
  Arms: TENS
Other: Physiotherapy technique: Vojta Therapy
  Arms: Vojta

SUMMARY:
This pilot "pre-post" quasi-experimental study evaluates for the first time the effectiveness of Vojta Therapy in treating lumbosciatic and compares it with the transcutaneous electrical nerve stimulation (TENS) procedure. Patients who agree will be distributed alternately in order of arrival to a Physiotherapy Unit, in such a way that half of the sample will be treated using TENS and the other half with Vojta.

DETAILED DESCRIPTION:
Lumbago/lumbosciatic (with or without radicular implication) is the second most frequent cause of primary medical care and the highest cause of disability in the entire world. This pathology is normally slight to moderate in the majority of cases, meaning that the therapeutical treatment tends to be conservative and thus the interest in increasing the range of non-invasive therapeutic possibilities is available.

Reflex Locomotion or Vojta Therapy began being used in 1959 for the rehabilitation of children with motor alterations and infants with a risk of cerebral palsy. Years later it was successfully applied to adults with neurological and motor alteration problems. Until now, there have been no studies on its use in pathologies of the spine and, in particular at a lumbar level.

A pre-/ post-intervention examination will be performed to obtain an objective clinical analysis (measurements of pain, disability, functionality and joint movement), by means of simple questionnaires completed by the patient (VAS scale, Oswestry and Roland-Morris questionnaires) and exploration techniques (Lasègue manoeuvre, Schöber test, fingertips to floor test and walking on heels and toes).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute, sub-acute or chronic lumbosciatic by a rehabilitation doctor were referred by said doctor to the Physiotherapy Unit, as candidates for either of the therapeutical procedures.

Exclusion Criteria:

* Patients with lumbosciatic resulting from a specific pathology (infection, metastasis, neoplasia, osteoporosis, fracture or inflammatory arthropathy).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Pain | 1 year
  To quantify pain, the investigators used two aggregated measures coming independently from the Visual Analogical Scale (VAS) and the Oswestry questionnaire.
  The Oswestry questionnaire has a scale both for back pain and for lower leg pain.
  VAS measures the intensity of pain subjectively described by the patient, with maximum reproducibility amongst observers. It consists in a graduated scale from 0 cm (extreme "no pain") to 10 cm (extreme "unbearable pain"), in which the patient establishes the point on the scale that best describes the intensity of the pain. It is universally used and relates well to descriptive scales, with good sensitivity and reliability

SECONDARY OUTCOMES:
Disability | 1 year
  To measure the degree of disability the investigators used two aggregated measures coming independently from the Oswestry and Roland-Morris questionnaires (validated Spanish versions).
  The Oswestry disability back pain questionnaire or Oswestry Disability Index (ODI), contains 10 items with 6 possible answers (0-1-2-3-4-5), from lowest to highest limitation. A clinically significant change was considered when improvement was at least 10%. It has a predictive value of the chronic degree of pain, duration of sick leave and resulting treatment. This scale is included in the highest level of methodological quality (level A) and has a correlation coefficient of 0.92.
  The Roland-Morris questionnaire contains 24 questions relating to the patient's daily activities with a yes/no possible response. The final score is a punctuation from 0 to 24; the higher the score the greater the disability. Clinically relevant changes are considered with a difference of 2 to 5 points.
Flexibility | 1 year
  To evaluate the ability of bending the spine (or degree of restriction), the investigators used two aggregated measures coming independently from the Schöber Test and Fingertips to Floor Test.
  Schöber Test: in a standing position, the L5 spinous process is located and marked. Then investigators then measure a distance of 10 cm towards the head and make another mark. The person is then asked to flex their torso and the length between both marks is recorded.
  Fingertips to floor (FTF) test: the person stands with straight knees and feet separated to waist level. In this position, participants are asked to bend over as far as possible and the distance reached is measured.
Radiculopathy | 1 year
  to determine the existence of sciatic nerve compression, the investigators used the Lasègue manoeuvre. Whilst lying down, the patient lifts their leg with the knee straight. It is a positive sign if the leg hurts at an angle from 30-70º. To determine whether the damaged nerve root is L5 or S1 (motor weakness), the investigators analysed the patient walking on their heels and toes. If the most affected nerve root was L5, the patient had difficulty walking on their heels. If the difficulty is walking on their tiptoes, it was S1.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Juarez, Principal Investigator — SESCAM